CLINICAL TRIAL: NCT03921463
Title: the Key Laboratory of Female Pelvic Floor Disorders Diseases, Beijing, China
Brief Title: Changes of Pelvic Floor Functions in Women at Different Postpartum Time
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH4
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- caesarean section
- vaginal delivery

INTERVENTIONS:
Other:  — This is an observational study

SUMMARY:
The main purpose of this study was to observe the pelvic floor muscle strength abnormalities of cesarean section and vaginal delivery at different time points within six months after delivery without any intervention. It was a prospective observational study, and the main study population was healthy postpartum women. Regular follow-up was conducted at 6 weeks, 9 weeks, 3 months, 4 months, 5 months and 6 months postpartum. The follow-ups included gynecological examination, pelvic floor electrophysiological indexes (category I and II muscle fiber strength and fatigue), questionnaire (ICI- Q-SF, OABSS, UDI-6), and pelvic floor ultrasound. The incidence of pelvic floor muscle strength abnormality at different postpartum time points was statistically analyzed, the high-risk factors of postpartum pelvic floor function abnormality caused by pregnancy and delivery were analyzed, and the general rules of the natural development of pelvic floor function were observed.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age: 20 ~35 years old; 2) first parturients registered in the obstetrics department of our hospital; 3) no medical complications before pregnancy, no UI and POP (according to the standard of POP-Q stage); 4) no obstetric complications; 5) the patients agreed to conduct the study and signed the informed consent.

Exclusion Criteria:

* 1) patients with uncontrolled epilepsy, central nervous system diseases or mental disorders, whose clinical severity shall be determined by the researcher to affect clinical research compliance; 2) follow up the patients with difficulty.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: healthy postpartum women
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of pelvic floor muscle strength abnormality at different postpartum time | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- The Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 month